CLINICAL TRIAL: NCT02978690
Title: Multi-centre, Open-label, Single Arm, Phase I Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacogenomics and Efficacy of a Single Intravenous Dose of Spesolimab in Patients With Active Generalized Pustular Psoriasis
Brief Title: Spesolimab (BI 655130) Single Dose in Generalized Pustular Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368.11; 2016-001236-35 (EudraCT Number)
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spesolimab (Experimental)
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Solution for infusion
  Other Names: BI 655130

SUMMARY:
This is a phase I, open label, single group study that is being performed to assess the safety, tolerability, Pharmacokinetics (PK) , Pharmacogenomics (PGx) and efficacy of a single dose of spesolimab in adult patients with active Generalized Pustular Psoriasis (GPP).

ELIGIBILITY:
Inclusion criteria:

* Male or female patients, aged 18 to 75 years at screening,
* A known and documented history of Generalized Pustular Psoriasis
* Presenting with a flare of Generalized Pustular Psoriasis
* A Generalized Pustular Psoriasis Physician Global Assessment score of at least moderate severity,
* Generalized Pustular Psoriasis patients receiving maintenance treatment with retinoids and/or methotrexate for at least 4 weeks or Generalized Pustular Psoriasis patients not receiving any maintenance therapy, at screening,
* Signed and dated written informed consent prior to admission to the study,
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

Male patients must be ready and able to use condoms.

- Further inclusion criteria apply

Exclusion criteria:

* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Immediate life-threatening flare of Generalized Pustular Psoriasis or requiring intensive care treatment, according, to the judgement of the investigator. Life-threatening complications mainly include, but are not limited to, cardiovascular/cytokine driven shock, pulmonary distress,
* Identified, ongoing serious/severe infection,
* Acute generalized exanthematous pustulosis (AEGP)
* Patient's clinical presentation being considered due to the differential diagnosis of toxic epidermal necrosis or Stevens-Johnson syndrome,
* Currently involved in or intending to participate in another investigational study during the course of this trial,
* Previous enrolment in this trial
* Use of any restricted medication, or any drug considered likely to interfere with the safe conduct of the study
* Background therapy with ciclosporin within the last 30 days preceding the second screening visit,
* Severe, progressive, or uncontrolled renal, hepatic, haematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms thereof, as judged by the investigator.
* Known chronic or relevant acute infections including active tuberculosis, HIV or viral hepatitis; QuantiFERON® tuberculosis test will be performed at screening. If the result is positive, patients may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment should have been initiated and maintained according to local country guidelines.
* Patient with a transplanted organ (with exception of a corneal transplant > 12 weeks prior to screening) or who have ever received stem cell therapy (e.g., Prochymal).

Known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.

* Any documented active or suspected malignancy or history of malignancy within 5 years prior to second screening visit, except appropriately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse) other than Generalized Pustular Psoriasis, surgical procedure (i.e., organ transplant), medical examination finding (including vital signs and electrocardiogram), or laboratory value at the second screening visit outside the reference range, that is in the opinion of the investigator, is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data,
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- HOP Saint-Louis, Paris, France
- Nagoya City University Hospital, Aichi, Nagoya, Japan
- Hospital Sultanah Aminah, Johor Bahru, Malaysia
- Pusan National Univ. Hosp, Busan, South Korea
- National Taiwan University Hospital, Taipei, Taiwan
- Hedi Chaker Hospital, Department of Dermatology, Tunisia, Tunisia

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Gwillim EC, Nichols AJ. Spesolimab for generalized pustular psoriasis: a review of two key clinical trials supporting initial US regulatory approval. Front Immunol. 2024 Jul 22;15:1359481. doi: 10.3389/fimmu.2024.1359481. eCollection 2024. PMID 39104539
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the screening visit, patients had to be on stable maintenance treatment (for at least 4 weeks) with retinoids and/or methotrexate or not to receive any maintenance therapy at all. All patients were to use an effective birth control method throughout the trial.
Pre-assignment Details: This exploratory, Phase I, multi-centre, multi-national trial in male and female patients with a flare of Generalised Pustular Psoriasis (GPP) applied an open-label design.
Groups:
- Spesolimab: Patients received a single intravenous dose of 10 milligram/kilogram (mg/kg) body weight spesolimab (BI 655130) in an open label manner.
  The intravenous infusion over 60 minutes (min), could be prolonged by the investigator up to 240 min.
  Patients were to be followed up for 140 days (20 weeks) after dosing.
Period: Overall Study
Arm/Group | Spesolimab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All patients in the treated set (TS) who had a baseline and at least one post baseline GPP Area and Severity Index (GPPASI) or GPP Physician Global Assessment (GPPGA) measurement and no important protocol violation flagged for exclusion from the FAS.
Arm/Group | Spesolimab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Reactions, Defined as Drug-related Adverse Events (AE)
Description: Percentage of patients with adverse reactions, defined as drug-related Adverse Events is presented.
Time Frame: Up to 140 days from the administration of spesolimab.
Population: Treated Set (TS): All patients who entered the trial and received the trial medication on Day 1 (Visit 3).
Measure: Number; unit: percentage of participants
Arm/Group | Spesolimab
Number analyzed (Participants) | 7
percentage of participants | 57.1

2. Secondary Outcome: Percent Change From Baseline in Generalized Pustular Psoriasis Area and Severity Index (GPPASI) Total Score at Week 2
Description: The GPPASI is an adaptation for Generalized Pustular Psoriasis (GPP) patients of the Psoriasis Area and Severity Index (PASI), an established measure of severity and area of psoriatic lesions in patients with psoriasis. It is a tool which provides a numeric scoring for patients overall GPP disease state, ranging from 0 (no disease) to 72 (worse disease state). It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, pustules, and scaling (desquamation) over four body regions. % GPPASI change from baseline=100* (GPPASI at baseline - GPPASI at post-baseline visit)/(GPPASI at baseline). For %GPPASI change, positive numbers show reduction in GPPASI with higher values representing a larger improvement or recovery of disease, while negative numbers show an increase in GPPASI, i.e. worsening of disease.
Time Frame: At baseline and at Week 2.
Population: Full Analysis Set Last Observation Carry forward (FAS LOCF). Full Analysis Set (FAS): All patients in the treated set (TS) who had a baseline and at least one post baseline GPP Area and Severity Index (GPPASI) or GPP Physician Global Assessment (GPPGA) measurement and no important protocol violation flagged for exclusion from the FAS. LOCF: The last available value, including baseline, was carried forward to all subsequent visits within the on-treatment period at which a measurement was missing.
Measure: Mean (Standard Deviation); unit: percent GPPASI change
Arm/Group | Spesolimab
Number analyzed (Participants) | 7
percent GPPASI change | 73.2 (16.2)

3. Secondary Outcome: Proportion of Patients With Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) Total Score of 0 (Clear) or 1 (Almost Clear) at Week 2
Description: GPPGA relies on clinical assessment of the GPP patient's skin presentation. It is a modified Physician Global Assessment (PGA), a physician's assessment of psoriatic lesions, which has been adapted to the evaluation of GPP patients.
  The investigator (or qualified site personnel) scores the erythema, pustules and scaling of all psoriatic lesions from 0 - 4. Each component is graded separately, the average is calculated and the final GPPGA is determined from this composite score. A lower score then indicates a lesser severity, with 0 being clear and 1 being almost clear. To receive a score of 0 or 1, the patient should be afebrile, in addition to skin presentation requirements.
Time Frame: At Week 2.
Population: Full Analysis Set No Response Imputed (FAS NRI). Full Analysis Set (FAS): All patients in the treated set (TS) who had a baseline and at least one post baseline GPP Area and Severity Index (GPPASI) or GPP Physician Global Assessment (GPPGA) measurement and no important protocol violation flagged for exclusion from the FAS. NRI: If there were data at the visits both immediately before and immediately after the visit with a missing outcome, a failure to achieve response imputed.
Measure: Number; unit: proportion of patients
Arm/Group | Spesolimab
Number analyzed (Participants) | 7
proportion of patients | 0.714

4. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score at Week 2
Description: Change from baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue scale scale score at Week 2 is presented.
  The FACIT-Fatigue scale is a brief and reliable instrument for monitoring fatigue and its effects on patients. It is a comprehensive compilation of questions that measure health-related quality of life in patients with chronic illnesses. It comprises 13 questions, the responses to which are each recorded on a 5-point Likert scale. Scores range from 0 to 52, with lower scores representing greater fatigue, i.e. higher changes from baseline indicate higher improvement (compared to baseline)
Time Frame: At baseline and at Week 2.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spesolimab
Number analyzed (Participants) | 7
units on a scale | 12.3 (10.1)

5. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (VAS) Score at Week 2
Description: The pain VAS is a unidimensional measure of pain intensity. It is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 millimeters (mm) in length, anchored by word descriptors at each end ('no pain', 'very severe pain'). The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the 'no pain' anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity, i.e., a negative change from baseline indicates an improvement (compared to baseline).
Time Frame: At baseline and at Week 2.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spesolimab
Number analyzed (Participants) | 7
units on a scale | -45.9 (32.3)

6. Secondary Outcome: Area Under the Concentration-time Curve of Spesolimab in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of spesolimab in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: Within 1.5 hours (h) before and 0.5 h, 24 h, 48 h, 72 h, 96 h, 120 h, 144 h, 312 h, 480 h, 648 h, 1992 h, 3336 h after spesolimab administration.
Population: Pharmacokinetic (PK) parameter set (PKS): All patients in the treated set (TS) who provided at least one secondary PK endpoint not flagged for exclusion due to a protocol violation relevant to the evaluation of PK (to be decided no later than at the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (μg)·day/ milliliter (mL)
Arm/Group | Spesolimab
Number analyzed (Participants) | 6
microgram (μg)·day/ milliliter (mL) | 2350 (41.1)

7. Secondary Outcome: Maximum Measured Concentration of Spesolimab in Plasma (Cmax)
Description: Maximum measured concentration of spesolimab in plasma (Cmax) is reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (μg)/milliliter (mL)
Arm/Group | Spesolimab
Number analyzed (Participants) | 6
microgram (μg)/milliliter (mL) | 203 (11.1)

ADVERSE EVENTS:
Time Frame: Up to 140 days from the administration of spesolimab.
Description: Treated Set (TS): All patients who entered the trial and received the trial medication on Day 1 (Visit 3).
Arm/Group | Spesolimab
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab (N=7)
Eosinophilia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chills (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Pharyngitis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral tonsillitis (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
Skin fragility (Skin and subcutaneous tissue disorders) | 1
Skin striae (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The results should be interpreted with caution given the limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT02978690/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT02978690/SAP_001.pdf